CLINICAL TRIAL: NCT03736746
Title: Testing Feasibility of Motivational Interviewing for Patient-Reported Cancer Pain Goals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other)
Responsible Party: Principal Investigator, Olga Ehrlich, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-376
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Other Cancer
Keywords: Other Cancer
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivational Interviewing (Experimental): * Will entail two-to-four Motivational Interviewing sessions per participant
  * Will include a battery of questionnaires
  * Investigator-led discussion about the participant's pain experience which is focused on the participant reporting of functional pain goals (FPGs).
  * The investigator will elicit questions and goals that participants will be encouraged to discuss with their palliative care providers
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — An investigator-led discussion about the participant's pain experience which is focused on the participant reporting of functional pain goals (FPGs)

SUMMARY:
This research study is evaluating the acceptability and feasibility of using a cognitive behavioral intervention called Motivational Interviewing to help persons with pain from cancer set goals for managing that pain.

DETAILED DESCRIPTION:
This study is being conducted to evaluate a new way that clinicians can help identify the goals that cancer participants have for managing their pain. This new method uses discussion between a patient and a clinician, in this case a registered nurse, during which one or more goals may be set. At this time, there are no tested methods that clinicians can use for helping patients set these kinds of goals.

ELIGIBILITY:
Inclusion Criteria:

* At least 18-years of age
* Has an appointment with DFCI ambulatory palliative care service for cancer-related pain
* Can speak English

Exclusion Criteria:

-Diagnosis of delirium or other cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of Motivational Interviewing intervention | 1 year
  The proportion of enrolled participants completing at least one follow-up Motivational Interviewing session (at least two sessions total). The proportion of participants completing at least one follow-up intervention session will be estimated along with an exact 90% confidence interval.

SECONDARY OUTCOMES:
Motivational Interviewing intervention usage rate | 1 year
  The number of interventions sessions attended divided by the total possible number of interventions sessions reported as the sample mean.
Participant intervention acceptability | 1 year
  The Participant Experience Questionnaire, developed by the investigator, will be used to summarize overall patient-reported acceptability in this study. Summary measures of median/range and mean/SD for total categorical scores, the time in weeks from the initial to follow-up intervention visit, and the number of completed intervention sessions will be reported.
Attitudinal barriers to pain | 1 year
  Attitudinal barriers to pain management will be measured using the Barriers Questionnaire-II which measures four attitudinal realms with 27 self-rated questions about pain beliefs. The total score will be calculated at study entry and after the first follow-up visit and scores will be summarized (median/range, mean/SD). If additional sessions are completed, the scores will be plotted over time and trends will be explored with graphical methods.
Pain Self-Efficacy | 1 year
  Pain self-efficacy will be measured using the Pain Self-Efficacy Questionnaire in which participants rate their confidence in daily living activities despite pain using a Likert-type scale.The total score will be calculated at study entry and after the first follow-up visit and scores will be summarized (median/range, mean/SD). If additional sessions are completed, the scores will be plotted over time and trends will be explored with graphical methods.
Observed engagement in goals-setting | 1 year
  Observed engagement will be evaluated using the instrument developed by the investigator for this study in which discussions of behaviors indicating active goal setting will be tabulated and salient quotes will be extracted for dissemination. Categories are:
  1. pain as an obstacle
  2. what helped pain before
  3. life with controlled pain
  4. suggestions to control pain
  5. suggestions actually used
  6. help-seeking
Motivational Interviewing intervention fidelity | 1 year
  Fidelity to Motivational Interviewing methods will be assessed on 33% of interviews using the Motivational Interviewing Skills for Health Care Encounters which is used to evaluate the degree to which the person providing the intervention follows five domains key to Motivational Interviewing.The domains are:
  1. Motivational Interviewing philosophy
  2. health interviewing
  3. motivation
  4. Motivational Interviewing principles
  5. interpersonal process
  Each domain has specific behaviors that are rated as:
  1. deficient
  2. developing
  3. accomplished
  4. not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Olga Ehrlich, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03736746/Prot_SAP_000.pdf